CLINICAL TRIAL: NCT04498546
Title: The Effects of Mask Usage on Exercise Capacity and Related Parameters During the COVİD-19 Pandemic
Brief Title: Mask Usage and Exercise During the COVİD-19 Pandemic
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Büşra Alkan, Research Assistant, KTO Karatay University
Other Study IDs: KaratayU3
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Exercise Test
Keywords: exercise capacity; surgical mask; exercise test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the effect of using mask during exercise on exercise capacity and values measured before exercise (heart rate, blood pressure, peripheral oxygen saturation (SpO2), fatigue, severity of dyspnea, etc.). To investigate the haemodynamic effects (heart rate, blood pressure, peripheral oxygen saturation (SpO2), fatigue, dyspnea severity, etc.) of the mask, which entered daily life during the epidemic period and which requires long-term use, and examine the effect on hemodynamic stress.

DETAILED DESCRIPTION:
Surgical masks are frequently used after the necessity to use a mask in the community.The effects of technologically well-designed training masks used in athletes have been shown on hypoxia and heart rate responses during exercise, but there are no studies examining the exercise capacity and hemodynamic responses given to exercise in healthy normal individuals.This study is planned to evaluate the effects of the use of surgical masks that are widespread in the community due to pandemic on the exercise capacity and exercise responses (heart rate, blood pressure, peripheral oxygen saturation, fatigue).

Exercise tests will be carried out for each individual randomly, twice with a mask and without a mask. The materials used before and after each exercise test will be sterilized. During the exercise test, individual antibacterial filters will be used for each person.Bruce protocol will be used to determine exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to be included in the research,
* Being between the ages of 18-65,
* Having physical fitness to do exercise tests,
* Having a cognitive function that will allow active participation in the exercise test.
* No chronic illness.

Exclusion Criteria:

* Not to volunteer to participate in the research,
* Having any mental or physical condition that impedes performing exercise tests,
* Having any of the symptoms of COVID-19,
* Having been diagnosed with COVID-19 before,
* Having a history of contact with COVID-19 patient
* Having a cardiac, neurological, orthopedic and respiratory disease
* Use of assistive devices while walking

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers between the ages of 18-65 who are able to perform exercise tests will be included in the study.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Resting Heart Rate | baseline
  Resting Heart Rate beats/min
Peak Heart Rate | During the procedure
  Peak Heart Rate beats/min
Recovery Heart Rate | Immediately after the procedure
  Recovery Heart Rate beats/min
Resting systolic blood pressure | baseline
  Resting systolic blood pressure mmHg
Recovery systolic blood pressure | Immediately after the procedure
  Recovery systolic blood pressure mmHg
Resting diastolic blood pressure | Baseline
  Resting diastolic blood pressure mmHg
Recovery diastolic blood pressure | Immediately after the procedure
  Recovery diastolic blood pressure mmHg
Peripheral oxygen saturation | Baseline
  To be measured by Pulse Oximeter (SpO2) To be measured by Pulse Oximeter (SpO2)
Peripheral oxygen saturation | Immediately after the procedure
  To be measured by Pulse Oximeter (SpO2)
VO2max | Baseline
  Maximal Oxygen Consumption (ml/kg/dk). Gas analyzer measuring breath to breath will be used.

SECONDARY OUTCOMES:
Dyspnoea Severity | Baseline
  It will be measured with a 20-point borg scale. As the score increases, the severity of dyspnea increases
Dyspnoea Severity | Immediately after the procedure
  It will be measured with a 20-point borg scale. As the score increases, the severity of dyspnea increases

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Özalevli, Prof, PT, Study Director — Dokuz Eylul Univesity; Özlem Akkoyun Sert, Phd, PT, Study Chair — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

REFERENCES:
- [Derived] Alkan B, Ozalevli S, Akkoyun Sert O. Maximal exercise outcomes with a face mask: the effects of gender and age differences on cardiorespiratory responses. Ir J Med Sci. 2022 Oct;191(5):2231-2237. doi: 10.1007/s11845-021-02861-3. Epub 2021 Nov 26. PMID 34837141